CLINICAL TRIAL: NCT05884190
Title: Community-based, Family-centered, Trauma-informed Approach to Timely Detection and Management of Early Postpartum Hypertension
Brief Title: Trauma-informed Approach to Timely Detection and Management of Early Postpartum Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000033779; MMM-2021C2-23671 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Postpartum Hypertension

STUDY DESIGN:
Intervention Model Description: The study population will include adult postpartum women at least 18 yrs old that are at-risk for hypertension and/or poor mental health outcomes. This is a multi-site intervention study that follows a sequential stepped-wedge design with the 3 hospitals randomized to their start time for the first arm followed by the second and third arms.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (SoC) (Active Comparator): Standard of Care for Postpartum Hypertension
  Interventions: Other: SoC
- Remote Medical Model (RMM) (Experimental): Includes SoC plus RMM
  Interventions: Other: Remote Medical Model (RMM); Other: SoC
- Community Health Model (CHM) (Experimental): Includes SoC, RMM plus CHM
  Interventions: Other: Remote Medical Model (RMM); Other: Community Health Model (CHM); Other: SoC

INTERVENTIONS:
Other: Remote Medical Model (RMM) — Remote home blood pressure (BP) monitoring once a day for the first 7 days and then at least weekly or more frequently as per a standardized blood pressure protocol up to six weeks and weekly virtual visits for 6 weeks and up to 12 weeks as needed by a physician extender (e.g. Nurse Practitioner, Pharmacist, etc.), and screening for social determinants of health and anxiety/ depression with referral for services if positive
  Arms: Community Health Model (CHM); Remote Medical Model (RMM)
Other: Community Health Model (CHM) — Utilization of community health workers trained in a strength-based trauma informed dyadic evidence-based approach.
  Arms: Community Health Model (CHM)
Other: SoC — SoC for Postpartum Hypertension

SUMMARY:
The investigators primary project goal is to improve clinical outcomes, including mental health outcomes, among postpartum at-risk women experiencing health disparities by increasing awareness, detection, and timely care of postpartum hypertension, mental health and cardiovascular complications. The investigators will accomplish this by comparing the effectiveness of two multi-component multi-level healthcare delivery models focused on early detection and control of postpartum hypertension and the social and mental health factors known to impact maternal outcomes, with the current standard of care and with each other.

DETAILED DESCRIPTION:
This study will compare two interventions with the standard of care. Given that this is a stepped-wedge design, all sites will begin with recruitment for the standard of care. All study participants will be identified, recruited and enrolled during their postpartum hospital stay (i.e. prior to discharge) by research study staff. Once study participants are enrolled, they will receive a Omron blood pressure (BP) cuff and will be instructed on how to use it.

General Design Description Overall study design. This project spans three states (Connecticut, Massachusetts, New York) and includes three hospitals (Yale New Haven Hospital, UMass Worcester, and Oishei in Buffalo, New York). This is a multisite intervention study that follows a sequential stepped-wedge design with the 3 hospitals randomized to their start time for the first arm followed by the second and third arms.

Yale will serve as the coordinating center and facilitate as well as oversee the planning and implementation activities across sites to ensure standardization. All study staff at all centers will undergo training sessions in blood pressure measurement and management following a standardized protocol as well as mental health screening and management and refresher training sessions, as needed, including any remedial training in specific areas targeted by quality control monitoring for a specific site. Yale New Haven Hospital will provide the appropriate assistance across clinical sites. This may include site visits, to ensure that the study enrollment and treatment follows proper study procedures.

Community Advisory Boards (CABs) will be formed at each of the project sites to integrate community perspectives into project activities and ensure community engagement in the decision-making process throughout the duration of the project. The Yale Griffin Prevention Research Center (PRC) and Cicatelli Associates, Inc. (CAI) will be deeply engaged advising on the establishment of the CABs across sites. Twice a year, the three CABs will convene virtually to receive an update about the overall project progress and share ideas about strengthening study design and implementation to ensure it reflects overall community needs and best interests. We will compensate members for their participation and transportation plus provide refreshments for in-person meetings. During in-person meetings of the individual site CABs, current COVID protocols recommended by the Centers for Disease Control will be followed to ensure meetings are safe and participants protected.

This study will compare two interventions with the standard of care. Given that this is a stepped-wedge design, all sites will begin with recruitment for the standard of care. All study participants will be identified, recruited and enrolled during their postpartum hospital stay (i.e. prior to discharge) by research study staff. Once study participants are enrolled, they will receive a Omron blood pressure (BP) cuff and will be instructed on how to use it.

Participants in the first intervention RMM will be provided with an Omron blood pressure cuff and blood pressure data will be recorded. Participants will be contacted within 72 hours following discharge. Follow-up telehealth visits will occur at least 1 time per week for the first 6 weeks and up to 12 weeks as needed. There may be a need for more visits for those with high blood pressure or elevated scores on validated mental health screeners, therefore advanced practice professionals (APPs) will coordinate with the individual site team Co-Is to address and arrange for additional follow-up visits with the appropriate providers as indicated.

In addition to the RMM described above, the second intervention, the community health model (CHM), includes the incorporation of research community health workers(CHW)/doulas who will be identified at each site. The CHWs/doulas will receive extensive training to be able to provide postpartum hypertension support and how to engage individuals in mental health services using a strengths-based trauma-informed approach. CHWs/doulas will be available to the families during the first 6 weeks (at least 1x per week) and then every other month or as needed. A hybrid approach will be used with CHWs/doulas visiting participants in-person and virtual based on the participant's needs and preferences.

All participants will complete assessments and a blood pressure at intake along with telephone follow-up assessments at 6 weeks postpartum, 3 months and 6 months postpartum including a blood pressure check and mental health screen with EPDS and other study surveys at each time point. Electronic medical record data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Delivery of singleton live birth (twins reduced to singleton or with vanishing twin syndrome prior to 14 weeks qualify)
* Postpartum
* English or Spanish speaking
* Viable pregnancy 24 weeks of gestation or above (Child can be in NICU to participate)
* Medicaid or the equivalent within each state (for example, Connecticut has Husky insurance) or uninsured
* Must living in one of the three states involved in this study (Connecticut, Massachusetts, New York) and preferably within the geographical area of each of the hospitals

Exclusion Criteria:

* Multifetal pregnancy (since are they at increased risk for key outcomes)
* Gestational age <24 weeks;
* Known major fetal anomaly in current pregnancy or stillbirth
* Actively using illicit/illegal substances (such as cocaine, heroin and other types of illicit opiates such as fentanyl) as noted in delivery hospitalization notes
* Active suicidal ideation with intent and plan
* Known primary psychotic disorder (i.e. schizophrenia, or schizoaffective disorder)
* Plans to move out of the state within 6 months
* Incapable of consent
* Severe medical complications that don't allow a mother to do the study effectively (for example, active treatment for cancer, dialysis etc. )
* Physician or provider refusal
* Patient refusal
* Incarcerated or institutionalized
* Stillbirth

Births that result in the newborn being under the care of another person or institution other than the birthing individual (e.g. adoption, state involvement) will be evaluated on an individual basis to determine if that person should be included.

For participants without access to a phone, we will explore if there are options that will allow them to have access to a devise for the times when they need to communicate with the study team. If not, they will not be able to participate in the study since this study requires phone or telehealth communication with research staff and/or APPs, and CHWs depending on study phase.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6030 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change in mean postpartum systolic blood pressure (SBP) at 6 weeks | 6 weeks
  Change in mean postpartum systolic blood pressure (SBP) at 6 weeks. A reduction in SBP indicates an improvement in postpartum hypertension.
Depression severity at 3 months postpartum assessed using the Edinburgh Postnatal Depression Scale (EPDS). | 3 months
  EPDS is a 10-item validated scale that measures depressive symptoms and is designed for use with pregnant and postpartum women. Scoring: None or minimal depression (0-6), Mild depression (7-13), Moderate depression (14-19), Severe depression (19-30). A reduction in depression severity at 3 months postpartum indicates a positive outcome.

SECONDARY OUTCOMES:
Participant engagement | 6 weeks
  Engagement with a health care provider by 6 weeks will be assessed via self-report (collected via interview) and electronic medical records (indicator will be whether the participant was engaged in care at least once in the 6 weeks postpartum).

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Pérez-Escamilla, PhD, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Massachusetts Memorial Health, Worcester, Massachusetts
  - Oishei Children's Hospital University at Buffalo, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No